CLINICAL TRIAL: NCT00147849
Title: A Cluster Controlled Trial Comparing Three Methods of Disseminating Practice
Brief Title: A Cluster Controlled Trial Comparing Three Methods of Disseminating Practice Guidelines for Children With Croup
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Institutes of Health Research (CIHR) (Other Government)
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: MCT-63141; CIHR App No. 110642; U Calgary Acct. No. 73-1051
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2005-11-29 (Estimated); Status verified 2005-09

CONDITIONS: Croup
Keywords: knowledge translation; health care utilization; economic analysis
MeSH Terms: conditions — Croup; Patient Acceptance of Health Care

INTERVENTIONS:
Behavioral: mailing of printed educational materials
Behavioral: a combination of interactive educational meetings, educational outreach visits, and reminders
Behavioral: identification of local opinion leaders and establishment of local consensus processes

SUMMARY:
The purpose of this study is to identify, from a societal perspective, the costs and associated benefits of three strategies for disseminating and implementing a practice guideline that addresses the management of croup.

DETAILED DESCRIPTION:
Overall Aim: The overall aim of this study is to identify - from a societal perspective - the costs and associated benefits of three strategies for implementing a practice guideline that addresses the management of croup.

Intervention Strategies: The intervention strategies to be compared will be mailing of printed educational materials (the "Standard intervention"), mailing plus a combination of interactive educational meetings, educational outreach visits, and reminders (a "Saturn intervention"), and a combination of mailing, interactive sessions, outreach visits, reminders plus identification of local opinion leaders and establishment of local consensus processes (a "Cadillac intervention").

Primary Objective: To determine which of the three intervention strategies are most effective at lowering the rate of hospital days per 1,000 disease episodes. The null hypothesis is that none of the intervention strategies reduce hospital utilization rates from baseline. The alternate hypothesis is that the intervention strategies will have a graded degree of effect on hospitalization rates, with the 'Standard intervention' having minimal to no effect, the 'Saturn intervention' having moderate but significant effect, and the 'Cadillac intervention' having the greatest effect.

Secondary Objective: To determine which of the three dissemination strategies are most effective at increasing the use of therapies of known benefit.

Economic Analysis: To determine which of the three intervention strategies will most effectively reduce total societal costs including all health care costs, costs borne by the family, and costs stemming from the strategies for disseminating guidelines.

Other Objectives: To determine which dissemination strategy will most effectively maintain or improve clinical outcomes and maintain or reduce the family psychosocial burden. Clinical outcomes assessed will include both uncommon severe events such as endotracheal intubation, respiratory arrest, and death, as well as average duration of clinical symptoms. The assessment of family psychosocial burden will include the number of hours of sleep missed by the child, and the stress experienced by the primary caregiver (most commonly the mother).

Study Plan: The study objectives will be achieved through the following:

1. We are completing a baseline survey which a) documents Alberta-wide utilization rates for health care services; b) documents severe adverse outcomes Alberta-wide; c) rank orders Alberta hospitals based on rates of hospitalization; d) documents therapeutic practices in 24 selected Alberta hospitals; and e) documents, through the use of a prospectively administered survey, the psychosocial burden of the disease on families in the same 24 Alberta hospitals.
2. We are developing clinical guidelines that address indications for drug therapy and hospital admission/discharge criteria. Development of these guidelines have included the following: a)convening an expert panel; b) critically reviewing the published literature; c) drafting guidelines which meet standard criteria for developing guidelines; d) obtaining approval of the guidelines by the Canadian Pediatric Society, Canadian Association of Emergency Physicians, and the Alberta Medical Association; and e) publishing the guidelines in journals such as the CMAJ.
3. We have identified 24 Alberta hospitals and will randomize them to one of the three dissemination strategies outlined above.
4. We will complete a follow-up survey which a) documents Alberta-wide severe adverse outcomes and utilization rates; b) documents practice patterns in the same 24 Alberta hospitals surveyed at baseline; and c) documents the psychosocial burden of the disease on families in these same hospitals.
5. We will complete a statistical analysis comparing the three randomized groups of hospitals in terms of the change in health care utilization, change in physician use of effective therapies, and change in the psychosocial burden of the disease on families.
6. We will complete an economic analysis that compares the change in benefits derived from the three types of dissemination strategies with the relative costs (change in health care costs, relative costs associated with the three types of dissemination strategies, and change in costs borne by the family such as lost wages).

ELIGIBILITY:
Inclusion Criteria:

* Alberta hospitals were rank ordered based on the number of disease episodes and rates of hospitalization for a six-year period. We then approached in this order each of the hospital administrators and clinical staff for permission to include their hospital in our study until a total of 24 hospitals consented

Exclusion Criteria:

* Refusal by hospital staff to participate in this trial

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-09; Study Completion 2006-03

PRIMARY OUTCOMES:
Rate of hospital days per 1,000 disease episodes

SECONDARY OUTCOMES:
Proportion of patients treated in the ED and hospital with a corticosteroid.
Proportion of patients evaluated in ED for at least three hours after treatment with corticosteroids before the decision to admit to hospital is made.
Time to treatment with corticosteroids in both ED and hospital patients.
An economic analysis conducted from a societal perspective with costs classified as either payer (costs born by the province) or non-payer (costs born by individuals or the families of children with croup).

CONTACTS AND LOCATIONS:
Overall Officials: David W Johnson, MD, Principal Investigator — University of Calgary